CLINICAL TRIAL: NCT03795181
Title: Prediction Model for Multiple Pulmonary Nodules
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jun Wang, Chief，Thoracic Surgery Service, Peking University People's Hospital
Other Study IDs: PTHO1902
Record Dates: First submitted 2019-01-01; First posted 2019-01-07 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Multiple Pulmonary Nodules
Keywords: multiple pulmonary nodules; predictive model
MeSH Terms: conditions — Multiple Pulmonary Nodules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study compares the sensitivity, specificity and accuracy of radiologists, thoracic surgeons and a predictive model (PKUM model) to discriminate malignancy from benign nodules in patients with multiple pulmonary nodules.

DETAILED DESCRIPTION:
It is clinically difficult to diagnose and manage patients with multiple pulmonary nodules (MPNs). We have developed a web-based mathematic model (PKUM model) by using a multi-centric database from three institutions (Peking University People's Hospital, Haidian Section of Peking University Third Hospital, People's Hospital Affiliated to Hebei Medical University) to predict the probability of a nodule to be malignant in patients with MPNs. This prospectively observational study will recruit patients with MPNs between January 2019 and March 2019, allowing radiologists, surgeons, and a predictive model (PKUM model) to discriminate malignancy from benign nodules, and compare their sensitivity, specificity, and accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly discovered, 4-30 mm multiple pulmonary nodules shown on thoracic CT scans
* Patients with at least two nodules resected for pathological evaluation

Exclusion Criteria:

* History of malignancy within 5 years
* Presence of pneumonia or pleural effusion on thoracic CT scans
* Patients with none or only one nodule resected
* Patients with initial chemo-radiation therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population include patients with multiple pulmonary nodules who will be diagnosed and treated between January 1，2019 and March 30, 2019. Patients with at least 2 nodules resected will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Performance of PKUM model | 3 months
  Area under receiver operating characteristic curve (AUC) of PKUM model in predicting the probability of a nodule to be malignant in patients with multiple pulmonary nodules.

SECONDARY OUTCOMES:
Comparison between PKUM model and clinicians | 3 months
  Comparison of sensitivity and specificity of radiologists, thoracic surgeons, and PKUM model in predicting the probability of a nodule to be malignant in patients with multiple pulmonary nodules.
Performance of PKUM model in equivocal nodules which is difficult to judge by clinicians | 3 months
  Sensitivity and specificity of PKUM model in predicting malignant probability of equivocal nodules judged by radiologists and thoracic surgeons.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, Principal Investigator — Peking University People's Hospital; Yuqing Huang, Study Director — Haidian Section of Peking University Third Hospital; Jiabao Liu, Study Director — People's Hospital Affiliated to Hebei Medical University; Yingtai Chen, Study Director — Beijing Aerospace 711 Hospital; Mingru Li, Study Director — Beijing Aerospace 731 Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China